CLINICAL TRIAL: NCT03801577
Title: Hepaxa Management of Non-Alcoholic Fatty Liver Disease (NAFLD): A Real-world Pilot Study Observing Effects of Nutritional Management With Hepaxa in Subjects With Liver Steatosis
Brief Title: Hepaxa Management of Non-alcoholic Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BASF AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTN01019401
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non Alcoholic Fatty Liver; NASH - Nonalcoholic Steatohepatitis
Keywords: omega-3; nafld; nafl; nash; medical food
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Subjects are screened for eligibility and on consent, historical data from liver fat measurements With CAP scores, will be collected from the previous 6 months. Only subjects With no, or poor response to lifestyle recommendations will be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepaxa (Experimental): Subjects will receive Hepaxa according to standard use (4 capsules daily over a 6 month period)
  Interventions: Dietary Supplement: Hepaxa

INTERVENTIONS:
Dietary Supplement: Hepaxa — High concentrate EPA and DHA

SUMMARY:
This study measures the steatosis in patients With fatty livers as determined by CAP score from a fibroscan assessment. The study attempts to determine the effect of using the Medical Food Hepaxa in a Clinical setting Close to real-world use.

DETAILED DESCRIPTION:
Subjects With fatty liver are given Hepaxa for 6 months. Fibroscan CAP measurements are taken at 3 monthly intervals. Subjects consent to Collection of data from approximately 6 months prior to use of Hepaxa. Patients unresponsive to life style recommendations given as standard practice will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, ≥18 years of age.
2. Suspicion of NAFLD
3. Able to understand and cooperate with study procedures, and have signed a written informed consent prior to any study procedures.
4. CAP score at -6 months and at inclusion of >268
5. A fibroscan elastography score <9 Kpa (Advanced Fibrosis)

Exclusion Criteria:

1. Other causes of liver inflammation including Hepatitis A, B or C, HIV, confirmed or suspected cirrhosis, Wilson's disease, autoimmune hepatitis, hemochromatosis, alcoholic steatohepatitis, pancreatitis, or prescription medications known to cause liver damage, or known to be hepatotoxic.
2. Significant weight loss (> 5% body weight) or rapid weight loss (>1.6 kg/week), within six months of screening.
3. Individuals taking prescription or supplemental omega-3 fatty acids.
4. Has a condition the Investigator believes would interfere with the evaluation of the subject, or may put the subject at undue risk during the course of the study, including potentially abnormal lab results, due to a traumatic event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The change in liver fat content (hepatic steatosis) from baseline to end of study | 6 months
  Liver fat will be measured using the "Controlled Attenuation Parameter" from the ultrasound based Fibroscan machine

SECONDARY OUTCOMES:
Change in liver function test: aspartate aminotransferase (AST) from baseline (IU/L) to end of study | 6 months
  Blood test
Change in the liver function test: alanine aminotransferase (ALT) from baseline (IU/L) to end of study | 6 months
  Blood test
Change in the liver function test: gamma glutamyltransferase (GGT) from baseline (IU/L) to end of study | 6 months
  Blood test
Change in Level of plasma triglycerides from baseline to end of study | 6 months
  Blood test
Change in weight from baseline to end of study | 6 months
  Blood test

OTHER OUTCOMES:
Exploratory outcome. Stratification of effect Hepaxa using FLI score | 6 months
  The fatty liver index score will be used to stratify patients for analysis of effect of Hepaxa

CONTACTS AND LOCATIONS:
Overall Officials: Reed Hogan, MD, Principal Investigator — GI Associates and Endoscopy Center
Locations (1):
- GI Associates and Endoscopy Center, Flowood, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
Only anonymized data will be shared With the Sponsor. The study protocol and report may be shared, and presented as Scientific posters and peer-reviewed articles.